CLINICAL TRIAL: NCT05253924
Title: Biological Underpinnings of Socio-emotional Regulation in Preterm Infants and Healthy Controls: Insights From EEG and Epigenetic Data
Brief Title: Biological Underpinnings of Socio-emotional Regulation in Preterm Infants and Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: Id. 867
Record Dates: First submitted 2022-02-01; First posted 2022-02-24 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Preterm Birth; Parent-Child Relations; Epigenetics
Keywords: At-risk Infants; Developmental Care; DNA methylation; Affectionate touch; Frontal alpha asymmetry
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will investigate the methylation status of target genes (such as BDNF, SLC6A4, OXTR, NR3C, Piezo1, Piezo2, TRPV1 andTRPM8) in saliva samples of preterm children (PT), compared with a sample of full term children (FT). Saliva sample will be collected for both PT and FT groups. Saliva samples will be obtained by a trained researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm children (PT): gestational age at birth <37
  Interventions: Diagnostic Test: DNA methylation of target genes; Diagnostic Test: EEG acquisition
- Full-term children (FT): gestational age at birth ≥ 37 weeks
  Interventions: Diagnostic Test: DNA methylation of target genes; Diagnostic Test: EEG acquisition

INTERVENTIONS:
Diagnostic Test: DNA methylation of target genes — The methylation status of target genes (BDNF, SLC6A4, OXTR, NR3C1, Piezo1, Piezo2, TRPV1 andTRPM8) will be investigated. Saliva sample will be collected for PT and FT. Genomic DNA will be extracted from aliquots of 0. 4 ml of each saliva sample with the Oragene OG575 (DNA Genotek) and stored at -20°C. Aliquots of 250 ng of each DNA will be edited for methylation analysis with the EZ DNA Methylation Lightning kit (Zymo Research). Amplification of samples and their preparation for NGS sequencing will be performed. Samples will be sequenced on NextSeq 500 (Illumina). Individual processed sequences (PE reads) will be independently aligned to reference sequences using a parallel Smith-Waterman algorithm. Only reads that consistently align to the same reference sequence will be retained. At each CpG site in each analyzed sequence, the frequencies of the four bases will be evaluated.
Diagnostic Test: EEG acquisition — Both PT and FT infants will have their EEG signal recorded during mother-baby interaction according to a modified version of the Still Face paradigm; the EEG signal will be recorded by means of the medical system eego mylab (AntNeuro), using special headphones equipped with 32 electrodes and suitable to acquire the EEG signal since early childhood. After spectral analysis of the EEG signal, the difference in signal strength in the alpha band recorded by two homologous electrodes (or electrode clusters) (i.e. right alpha - left alpha) will be calculated to obtain the FAA index. Because the alpha frequency band is associated with cortical inhibitory activity, a lower asymmetry reflects less left hemisphere activation than right hemisphere activation. The analysis of EEG data will be performed in MatLab environment using the eeglab software and algorithms developed ad hoc.

SUMMARY:
Preterm infants (PT) often need to spend their first weeks of life in the Neonatal Intensive Care Unit (NICU) where they are exposed to several adverse conditions. Whereas a consistent number of studies suggest that NICU-related experiences may have effects on infant development including long-term impairments in emotional regulation, the underlying mechanisms remain partially unexplored. Spectral analysis of EEG signal has demonstrated that frontal alpha-band asymmetry represents a reliable biomarker of social-emotional functioning. In the literature, higher right frontal activation has been associated with worse emotional regulation but no study has measured this value during a condition of social-emotional stress such as the Still Face paradigm. Our hypothesis is that higher alpha activity will be recorded in right frontal areas in premature infants compared to healthy controls and that this activation will be associated with higher negative emotionality (i.e., worse socio-emotional regulation) expressed during the Still Face paradigm. Moreover, despite several changes in epigenetic patterns have already been reported in association with prematurity and early adverse experiences, the relationship between epigenetic changes and electroencephalographic patterns (i.e. frontal alpha asymmetry) remains unexplored. The investigators therefore expect to find associations between increased methylation levels of socio-emotional and stress related genes (i.e. SLC6A4, NR3C1, OXTR, Piezo1, Piezo2, TRPV1 and TRPM8) with spontaneous oscillations of neural activity at frontal sites measured by EEG (i.e. frontal alpha asymmetry). Finally, there is ample evidence that infant's socio-emotional regulation abilities are highly dependent on the behaviors of their caregivers. More recent studies have shown that behavior can be influenced by interoceptive awareness, i.e., the ability to perceive the physiological condition of one's body in this way and to represent one's internal states. Better interoceptive awareness is associated with better recognition of others' needs, more empathetic behaviors, and better emotional regulation. Therefore, with the present exploratory study, the investigators will compare the interceptive awareness of mothers of preterm infants with that of mothers of full-term infants by exploring possible associations of this dimension with the socio-emotional responses of preterm infants and healthy controls. The investigators expect that better socio-emotional regulation of infants is predicted by a higher level of interoceptive awareness in mothers, regardless of prematurity condition.

DETAILED DESCRIPTION:
The main objective of the present study is to:

1. explore frontal and parietal alpha EEG signal asymmetry in association with social-emotional regulation in a group of preterm infants aged 6-12 months (age corrected, CA).

   Secondary aims are:
2. the investigation of epigenetic correlates (methylation of target genes:(i.e. SLC6A4, NR3C1, OXTR, Piezo1, Piezo2, TRPV1 and TRPM8) associated with social-emotional regulation
3. the contribution of mother's interoceptive awareness (Heartbeat Counting Task index) in social-emotional regulation in a sample of premature infants aged 6-12 months (CA).

The study involves the following procedures:

* EEG signal recording and analysis (frontal alpha rhythm asymmetry; FAA) in PT and FT infants
* Video recording of mother-child interaction in accordance with a modified version of the Still Face paradigm.
* Collection of biological material (DNA)
* Assessment of mothers' interoceptive awareness via Heartbeat Counting Task

Significance and innovation:

To the best of our knowledge, no study has evaluated the association between (1) EEG signal asymmetry, (2) methylation patterns of candidate genes, (3) mothers' interoceptive awareness (Heartbeat Counting Task index), and socio-emotional regulation in premature infants during the first months of life.

The present study will integrate several biomarkers and observational data to better elucidate the role of electroencephalographic activation patterns, epigenetic variations, and mothers' interoceptive awareness in the socio-emotional regulation abilities of infants born prematurely. In addition, a particularly novel aspect of this study is the application of EEG signal recording during the Still Face paradigm. The measurement of the EEG signal during this paradigm could increase our knowledge with respect to the brain mechanisms underlying socio-emotional regulation in premature infants and in healthy control.

Moreover, the focus on parental bodily states might provide a new perspective suggesting that enteroceptive awareness may contribute to support caregiver's ability to understand (and respond to) the infant's signals and emotional states.

Impact:

This study is warranted to provide relevant insights for the biochemical and neurological underpinnings of socio-emotional development in preterm infants and will provide new evidence-base information for improving the quality of supportive interventions for preterm infants and caregivers in and outside the NICU. In addition, the identification of potential electroencephalographic patterns associated with emotional regulation in premature and term infants may prove to be a novel biomarker for the early detection of children at risk for emotional and behavioral problems.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for PT infants are:

• gestational age< 37weeks;

Inclusion criteria for FT infants are:

• gestational age ≥ 37weeks;

Inclusion criteria for mothers are:

* mothers of Italian nationality;
* mother over 18 years of age;
* mother with absence of manifest psychiatric and/or cognitive pathologies (must be previously diagnosed major psychiatric pathologies);
* non-addicted/no habitual use of psychotropic medications, drugs, alcohol no smoking;
* non-single-parent families.

Exclusion Criteria: refer to inclusion criteria

-

Ages: 6 Months to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants. Preterm infants infants will be pre-screened for medical status variables by the NICU neonatologists of different hospital in Lombardy. Following a letter outlining the general research, parents will be meet per person in NICU or contacted by telephone and asked to voluntarily participate. Full-term infants. Mothers and their infants will be enrolled during the prenatal/postnatal parenting course in different hospital and nursery school in Lombardy. Following a letter outlining the general research, parents will be contacted by telephone and asked to voluntarily participate.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-13 (Estimated)

PRIMARY OUTCOMES:
Negative emotionality assessed during the Still-Face Paradigm (FFSF). | Once, From 6 to 12 months (CA for prematurity) of infant's life
  Negative emotionality (withdrawn, protesting, complaining, being fussy or crying behaviors) will be assessed using the validated coding system Infant and Caregiver Engagement Phases - ICEP. Coders have to detect the presence or the absence of negative emotionality-related behaviors for each episode of FFSF. Then, a proportion index of negative emotionality will be obtained for each of the five episodes of FFSF dividing the total score of negative emotionality displayed in every FFSF episode for the actual length of the episode, resulting in five negative emotionality indexes. Higher indexes of negative emotionality are indicative of worse social emotional regulation.
Frontal Alpha Asymmetry (FAA) | Once, From 6 to 12 months (CA for prematurity) of infant's life
  Frontal Alpha Asymmetry (FAA) will be assessed by computing the difference in signal power in the alpha band recorded by two homologous electrodes (or electrode clusters) (i.e. right alpha - left alpha). The EEG signal will be recorded through the medical system eego mylab (AntNeuro), using special headphones equipped with 32 electrodes and suitable to acquire the EEG signal since early childhood.
  Frontal Alpha Asymmetry (FAA) will also be correlated with Negative emotionality indexes.

SECONDARY OUTCOMES:
DNA methylation level of target genes | Once, From 6 to 12 months (CA for prematurity) of infant's life
  DNA methylation level of target genes will be assessed by the collection of a saliva sample using non-invasive modalities and the Oragene OG575 kit (Genotek DNA). Genomic DNA will be extracted, quantified with Qubit 2.0 (Invitrogen) and stored at -20°C at the Molecular Biology laboratory of the Scientific Institute E. Medea. Samples will be sequenced with NextSeq 500 (Illumina).
  DNA methylation levels of target genes will also be correlated with Negative emotionality indexes.
Heartbeat Counting Task index | Once, From 6 to 12 months (CA for prematurity) of infant's life
  Maternal perceptions of bodily self assessed by the Heartbeat Counting Task index.
  During the Heartbeat Counting Task mothers will be asked to mentally count the number of their own heartbeats over a period of time. The response will be compared with a measurement made using a pulse oximeter that allows for noninvasive determination of heart rate by photoplethysmography. The procedure is repeated in 4 different time intervals administered in random order among participants, without giving feedback on whether or not the responses are correct.
  Maternal perceptions of bodily self will also be correlated with Negative emotionality indexes.

CONTACTS AND LOCATIONS:
Locations (1):
- Associalzione La Nostra Famiglia - IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy